CLINICAL TRIAL: NCT06823869
Title: The Effect of Distraction Methods on Children Aged 3-6 Years Receiving Inhaler Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Berna Sözen, Nurse, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OndkusMU-SBF-BS-01
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Respiration Disorders
MeSH Terms: conditions — Respiration Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: this is a randoized controlled trial with a parallel assisnent design. participants will be randoly assgnrf to one of three groups: musical piano group, musical book group and control group (standard inhaler medication group). During the inhaler drug intake process, the child's fear and anxiety level will be compared between the three groups using distraction techniques.
Masking Description: ın this study , both the participants and the investigators are aware of the intervention being applied. participants in the musical piano group, musical book group and control group are informed about the specific treatment they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- musical book group (Active Comparator): During the inhaler medication treatment, the child will be accompanied by a toy doll with a nebul mask attached to its mouth, and the child will be asked which toy he would like to play with during the procedure. Children who answer musical books will be in this group.
  Interventions: Other: musical book
- musical piano group (Active Comparator): During the inhaler medication treatment, the child will be accompanied by a toy doll with a nebul mask attached to its mouth, and the child will be asked which toy he or she would like to play with during the procedure. Children who answer musical piano will be included in this group.
  Interventions: Other: musical piano
- group without toys (Sham Comparator): Children will not be given toys, and the researcher will show the child how to apply the inhaler medication on herself with a nebul mask before the treatment.
  Interventions: Other: sham

INTERVENTIONS:
Other: musical book — The child will indicate that he wants to play with the musical book. The child will play with toys for 5 minutes before treatment. Once the child is ready, inhaler medication will begin and the treatment will last 10 minutes. The treatment is terminated at the end of the 10th minute. The child's playing time with the toy is approximately 15 minutes.
  Arms: musical book group
Other: musical piano — The child will indicate that he wants to play with the musical piano. The child will play with toys for 5 minutes before treatment. Once the child is ready, inhaler medication will begin and the treatment will last 10 minutes. The treatment is terminated at the end of the 10th minute. The child's playing time with the toy is approximately 15 minutes.
  Arms: musical piano group
Other: sham — The child will not play with toys during treatment. Before the treatment, the researcher demonstrates the process on himself with a nebul mask. Treatment begins after the child is ready. The process will take 10 minutes.
  Arms: group without toys

SUMMARY:
The aim of this study is to observe the effect of distraction methods on children aged 3-6 years who apply to the emergency department due to respiratory complaints and receive inhaler medication.

DETAILED DESCRIPTION:
The research was designed based on voluntary participation in threegroups: the experimental group (doll and musical keyboard or musical book) and the control group. The inhaler drug application process is planned to be 10 minutes.

First, routine explanations are given to the children in the experimental group, and the child is ensured to be in an upright position for the parent to be present and to administer the inhaler medication. The child is explained that a doll will accompany him during the inhaler medication administration, and a nebulization mask is attached to the doll. Before starting the inhaler medication administration, the doll is placed next to the child in a sitting position. The child is asked to sit with the doll for 5 minutes and the child is asked whether he/she will play with a musical book or a musical piano.After the child decides which toy he/she will play with and plays with the toy for 5 minutes, the Child Fear Scale (CCS) and the Children's Emotional Indicators Scale (ÇEGÖ) are evaluated by the child, parent, researcher, nurse and vital signs before starting the procedure. Later, when the researcher decides that the child is ready for the procedure, inhaler medication administration is started. After the drug administration is completed, the child, parent, researcher and nurse evaluate the CQS and CEGRS, and vital signs are evaluated by the researcher, and the parent gives a parental satisfaction score.

In the control group, a routine explanation of the emergency department is given to the child and the parent, the parent is next to the child and the child is ensured to sit upright during the inhaler medication administration. To the children in the control group, the researcher shows how the procedure will be done with a nebula mask on himself. The procedure begins after the necessary explanations are made and the researcher decides that the child is ready for inhaler medication administration. Before starting the procedure, the child, parent, researcher, nurse and vital signs are evaluated by the researcher. After the inhaler intake is completed, ÇÖS and ÇEGÖ child, researcher, nurse, parent; Vital signs are evaluated by the researcher and parental satisfaction score is given by the parent.

ELIGIBILITY:
Inclusion Criteria:

* people who volunteer
* Children between 3 and 6 years old
* children without mental problems Children presenting to the emergency department with respiratory illnesses

Exclusion Criteria:

* children with a mental problem
* non-volunteers

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
child fear scale | 5 minutes before the intervention, during the process and just after the intervention was completed. 20 minutes in total.
  Child Fear Scale:It is used to measure the child's anxiety level. It ranges from neutral expression (0=no anxiety).
  A scale ranging from 0 to 4, consisting of five drawn facial expressions ranging from a scared face (4=severe anxiety).
  is the scale
Emotional Indicators Scale in Children | 5 minutes before the intervention, during the process and just after the intervention was completed. 20 minutes in total.
  It was developed by Ho Cheung, William Li and Violeta Lopez in 2005. In the scale, emotional indicators are evaluated according to 5 parameters. These parameters; facial expression, voice, activity, interaction and cooperation level. These five parameters are from 1 to 5.
  The lowest score in total is "5" and the highest score is "25".

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Esra Tural Büyük, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Samsun Ayvacık State Hospital, Ayvacık, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want my data to be used